CLINICAL TRIAL: NCT02474251
Title: Brain Sleep Clearance of Amyloid-Beta Peptides
Acronym: Brain SCRAPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-01837; 5R21AG049348-02 (NIH)
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Obstructive Sleep Apnea; Alzheimer's Disease
MeSH Terms: conditions — Sleep Apnea, Obstructive; Alzheimer Disease

STUDY DESIGN:
Masking Description: Mechanistic or physiologic study in humans.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): 25 cognitively normal elderly subjects (age 55-75), newly enrolled or currently participating in R01HL118624-01 (IRB S12-03068), a 2-year longitudinal on-going study that is aimed at examining the longitudinal associations between SDB and cognitive decline in the elderly.
  Interventions: Other: Continuous positive airway pressure device
- Group B (Active Comparator): 20 cognitively normal adults (age 30-75) with severe SDB (Apnea Hypopnea index [AHI]-all >30/hour) and good CPAP compliance from Mt. Sinai School of Medicnie (MSSM)
  Interventions: Other: Continuous positive airway pressure device

INTERVENTIONS:
Other: Continuous positive airway pressure device — GROUP B ONLY will be evaluated on two randomized counterbalanced nights, on one they will undergo a full night of therapeutic CPAP; on the other the investigators will withdraw CPAP during SWS only. A morning LP will be performed approximately 10 hours after sleep onset in both visits
  Other Names: CPAP

SUMMARY:
The 'Amyloid Cascade Hypothesis' posits that the accumulation of a peptide, amyloid beta (Aβ), in the brain is the initiating event in Alzheimer's disease (AD), however, the mechanisms involved are not well understood. Recent studies support the hypothesis that Aβ dynamics in the brain are influenced by the sleep-wake cycle, with increases in the production of soluble Aβ during wakefulness and decreases during non-rapid eye movement (NREM) sleep, and more specifically on NREM stage 3 (also called slow wave sleep [SWS]). These changes produce a consistent diurnal pattern in the cerebrospinal fluid (CSF) that has been documented in murine models and in humans. By better understanding this sleep-wake relationship the investigators hope to identify how sleep disorders accelerate the progression of AD in the elderly (which has been demonstrated by multiple epidemiological studies) and, in turn, identify novel therapeutic targets for AD prevention.

The purpose of this study is to elucidate how soluble amyloid beta (Aβ) levels in the brain are influenced by the sleep-wake cycle in humans, and to test the directionality of this relationship through sleep disruption experiments. The investigators will test two models. The first model will test how, prior to amyloid deposition, brain soluble Aβ levels may be relatively increased in the elderly by two mechanisms: a) loss of total sleep time and SWS that occur with normal aging; and b) sleep disturbances such as Sleep Disordered Breathing (SDB) or insomnia that are common in late life (Aim 1). The second model will test how stage-specific sleep disruption may lead to increased CSF Aβ42 levels (Aim 2). A group of adults with diagnosed severe SDB and good continuous positive airway pressure (CPAP) compliance will be used to test this model sleep deprivation experiments using therapeutic CPAP vs. sham CPAP.

This project will be the first to explore the protective effect of SWS on Aβ42 dynamics in a group of cognitively normal elderly subjects as well as the effect of acute sleep disruption by CPAP withdrawal on CSF Aβ42 levels in a well characterized clinical sample of severe obstructive SDB patients on treatment with CPAP. The results from this study will improve our understanding of the nature of the Aβ diurnal pattern and the brain consequences of full night sleep disruptions as well as sleep disruptions during specific stages of sleep.

DETAILED DESCRIPTION:
Evaluations and procedures performed by the participants in:

Aim 1 Subjects were newly enrolled normal elderly or normal elderly recruited from R01HL118624-01 and evaluated according to the studies protocol.

Visit 1: During this visit, participants will undergo a complete physical exam, neurological examination, psychiatric interview, sleep interview, neuropsychological testing, Heart testing (EKG), laboratory analysis of blood. (90cc)

Visit 2: During this visit, participants will undergo an MRI scan and be educated on completing home monitoring of sleep wake cycle with actigraphy.

Visit 3: Patients will receive one FBB PET/MR scan to establish amyloid status.

Visit 4: Patients will undergo one night of NPSG with maze task prior to the subjects' scheduled morning LP with collection of CSF (15 cc).

Aim 2 All subjects will receive a complete evaluation (outlined below). Visit 1 and visit 2 will be used to screen subjects for inclusion.

Visit 1: During this visit participant will undergo a complete physical exam, neurological examination, psychiatric interview, sleep interview, psychometric testing, heart testing (EKG), laboratory analysis of blood. (90cc)

Visit 2: During this visit patient will undergo an MRI scan and be educated on completing home monitoring of sleep wake cycle with actigraphy.

Visit 3: Patients will undergo one night of NPSG at MSSM with either consistent use of CPAP or use of Sham CPAP to model discontinuation. Approximately, 10 hours after sleep onset participant will have a LP with collection of CSF. They will also complete 3D Visual Maze task the night of in lab assessment and the morning after, right before the LP (15 cc).

Visit 4: Patients will undergo one night of NSPG at MSSM with either consistent use of CPAP or use of Sham CPAP to model discontinuation. Approximately, 10 hours after sleep onset participant will have a LP with collection of CSF. They will also complete 3D Visual Maze task the night of in lab assessment and the morning after, right before the LP (15 cc)

Incidental findings from study procedures (except for CSF analyses and ApoE genotyping) will be communicated to study subjects by the Study Physician.

ELIGIBILITY:
Inclusion Criteria:

Group A:

* Male and female subjects with normal cognition and 55-75 years of age
* Newly recruited or recruited on the follow-up evaluation from an existing longitudinal cohort of 180 normal elderly already enrolled in an active study (R01HL118624-01).

Group B:

* Male and female subjects with normal cognition and 30-75 years of age
* Recruited from the MSSM where there are already studies ongoing aimed at determining the consequence of disrupting REM sleep via CPAP withdrawal on the consolidation of spatial navigational memory (PI. Dr. Varga).
* Previously diagnosed moderate-severe SDB patients and on active CPAP treatment.

Group A + B:

* All subjects will be within normal limits on neurological and psychiatric examinations.
* All subjects enrolled will have both a Clinical Dementia Rating (CDR)<0.5 and Global Deterioration Scale (GDS)<3 (i.e. cognitively normal).
* All subjects will have an informed family member or life partner interviewed to confirm the reliability of the subject interview.
* All subjects will agree to the MRI imaging, the lumbar puncture (s), apolipoprotein E (ApoE) genotyping and DNA banking.

B. Exclusion Criteria:

* Diagnosis of any brain disease or MRI evidence of brain damage including significant trauma, hydrocephalus, seizures, mental retardation or other serious neurological disorder (e.g. Parkinson's disease or other movement disorders). Persons with silent cortical infarcts will be excluded. White matter lesions will not be exclusions.
* History of brain tumor or contraindications for LP.
* Prior history of post-LP headache.
* Significant history of alcoholism or drug abuse.
* History of major psychiatric illness (e.g., schizophrenia, bipolar or life long history of major depression)
* Geriatric Depression Scale >7 (for subjects > 55 y/o) or Beck Depression Inventory >18 (for subjects <55 y/o)
* Current pregnancy or intent to become pregnant during the period of study.
* Evidence of clinically relevant and uncontrolled cardiac (unstable and untreated coronary or peripheral artery disease), pulmonary (ventilatory failure, Cheyne-Stokes breathing, severe and inadequately controlled arterial hypertension, acute upper respiratory infection), untreated hypothyroid or uncontrolled hematological conditions. Insulin dependent diabetes and/or history of treated hypertension are not exclusions. Normal subjects with current levels of HbA1c >5.9% or diabetics >7.0% and/or current blood pressure levels >140/90 mm Hg will be advised to seek referral.
* Physical impairment of such severity as to adversely affect the validity of psychological testing.
* Any prosthetic devices (e.g., pacemaker or surgical clips) that constitutes a hazard for MRI imaging.
* History of a first-degree family member with early onset AD (< age 60) dementia.
* Prior bariatric surgery within 6 months or are currently participating in a medical weight loss program.
* Irregular sleep-wake rhythms (based on one week at home monitoring with actigraphy)
* Inability to avoid the use of alcohol, caffeine during the 48h before the NPSG .
* Patients that are professional vehicle drivers or train operators, or patients that have had a previous motor vehicle accident related to sleepiness and cannot rest the day of the LP after the sleep deprivation experiment.
* Conditions that alter normal sleep patterns: Irregular sleep-wake rhythms (based on one week at home monitoring with actigraphy) or moderate to severe SDB (AHI4%>15 per hour) .
* Medications adversely affecting cognition or sleep will result in exclusion. The excluded medications include:

  * Narcotic analgesics (>2 doses per week).
  * Chronic use of medications with anticholinergic activity.
  * Anti-Parkinsonian medications (carbidopa/levodopa, amantadine, bromocriptine, pergolide, selegeline).
  * Others: amphetamines, amphetamine-like compounds, appetite suppressants, phenothiazines, reserpine, buspirone, clonidine, disulfiram, guanethidine, MAO inhibitors, theophylline, tricyclic antidepressants, salicylates, cholinesterase inhibitors and memantine.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
CSF Aβ42/Aβ40 levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Osorio, MD, Principal Investigator — NYU MEDICAL CENTER
Locations (2):
- United States (2):
  - Bellevue Hospital Center, New York, New York
  - NYU Langone Medical Center, New York, New York

REFERENCES:
- [Background] Hardy JA, Higgins GA. Alzheimer's disease: the amyloid cascade hypothesis. Science. 1992 Apr 10;256(5054):184-5. doi: 10.1126/science.1566067. No abstract available.
- [Background] Kang JE, Lim MM, Bateman RJ, Lee JJ, Smyth LP, Cirrito JR, Fujiki N, Nishino S, Holtzman DM. Amyloid-beta dynamics are regulated by orexin and the sleep-wake cycle. Science. 2009 Nov 13;326(5955):1005-7. doi: 10.1126/science.1180962. Epub 2009 Sep 24. PMID 19779148
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Lucey BP, Bateman RJ. Amyloid-beta diurnal pattern: possible role of sleep in Alzheimer's disease pathogenesis. Neurobiol Aging. 2014 Sep;35 Suppl 2:S29-34. doi: 10.1016/j.neurobiolaging.2014.03.035. Epub 2014 May 15. PMID 24910393
- [Background] Bayer-Carter JL, Green PS, Montine TJ, VanFossen B, Baker LD, Watson GS, Bonner LM, Callaghan M, Leverenz JB, Walter BK, Tsai E, Plymate SR, Postupna N, Wilkinson CW, Zhang J, Lampe J, Kahn SE, Craft S. Diet intervention and cerebrospinal fluid biomarkers in amnestic mild cognitive impairment. Arch Neurol. 2011 Jun;68(6):743-52. doi: 10.1001/archneurol.2011.125. PMID 21670398